CLINICAL TRIAL: NCT03143179
Title: Acute Hemodynamic and Cardiac Responses to Spinal Cord Injury: A Feasibility Study
Brief Title: Acute Cardiac Responses to Spinal Cord Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Christopher West, Principal Investigator, University of British Columbia
Other Study IDs: H16-00818
Record Dates: First submitted 2017-05-02; First posted 2017-05-08 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The immediate period after spinal cord injury (SCI) is one of the only opportunities that clinicians and care-givers have to make a real difference to patient outcomes. One of the main aims during this period is to preserve blood flow and oxygen delivery to the spinal cord to prevent any further damage from occurring after the injury. The heart acts as the major pump for blood to be pumped to the spinal cord and the body. It has been shown in small animal models and in humans with long-standing SCI that the ability of the heart to pump blood after injury is compromised, which may in turn reduce the amount of blood and oxygen delivered to the injured cord. It is unclear how quickly these changes occur in the heart following SCI and how best to manage heart function such that blood flow and oxygen delivery can be optimized. In the present study, the investigators will examine how the heart functions immediately after SCI. The findings from this study are expected to provide new information that could help clinicians improve the management of people who have just suffered a SCI.

DETAILED DESCRIPTION:
Background:

The hemodynamic management of the cervical/high-thoracic spinal cord injured patient represents a remarkably complex clinical scenario, but represents one of the only potentially neuroprotective therapeutic options currently available to the clinician. Presently, the singular goal of hemodynamic management is to increase mean arterial blood pressure (MAP) to 85mmHg by targeting peripheral tone via vasopressor therapy, with a view to increasing perfusion of the spinal cord, preventing ischemia at the injury site, and optimizing neurological outcome. It is often overlooked that the instantaneous removal of descending sympathetic control at the time of SCI renders not only the vast majority of the systemic vasculature devoid of supraspinal input, but it also impairs descending control of the heart. What is yet to be considered in current hemodynamic management protocols is that immediate cardiac dysfunction secondary to impaired supraspinal control of the heart may very well be a significant contributor to poor spinal cord perfusion. Indeed, data collected over the last four years in rodent SCI models suggests that cardiac sympathetic decentralization is the principal cause of the low cardiac output observed in both rodents and people with chronic SCI. As such, the investigator's initiative is to provide a novel approach to hemodynamic management to a porcine model that harnesses both peripheral tone and cardiac function. The investigators believe this approach is an immediately translatable neuroprotective strategy for acute SCI.

Overview:

10 individuals aged 18-60 who have sustained an acute traumatic SCI (above T2 spinal level) less than 72 hours prior will be recruited over a period of 2 years. Recruitment will be isolated to those individuals who already have a central venous catheter and arterial line as part of standard clinical care (which actually occurs in most patients). In addition to standard clinical lines, an esophageal Doppler probe will be placed to measure aortic outflow on which beat-by-beat systolic cardiac function (i.e., stroke volume, cardiac output, ejection fraction) can be estimated. During a 120 min monitoring period, beat-by-beat dependent cardiac indices will be recorded and a modified Starling curve will be constructed by examining relationships between central venous pressure (i.e., an index of venous return) and aortic flow (i.e., an index of cardiac output). After 1hr of monitoring (Part A), a 250ml bolus of intravenous crystalloid will be infused over a 5 min period and measure beat-by-beat central venous pressure and aortic flow (stroke volume) responses (Part B). The primary outcomes are daily resting stroke volume and ejection fraction, change in stroke volume and central venous pressure (CVP) in response to fluid challenge. The secondary outcome is the slope of the Starling curve

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged 18-60yrs
* Acute traumatic SCI at T2 or above within the last 72 hours
* Complete (American Spinal Injuries Association Impairment Scale (AIS) A) or incomplete (AIS B) initial designation
* Requires insertion of central venous catheter and arterial catheter as part of standard clinical care
* Able to communicate in English and provide informed consent
* in sinus rhythm.

Exclusion Criteria:

* History and/or symptoms of cardiovascular disease or cardiopulmonary problems/disease, including controlled/uncontrolled hypertension
* Historical or current nasal injury (incl. cosmetic surgery)
* Nasal polyps
* Concurrent facial trauma
* Traumatic brain injury
* Concurrent intra-aortic balloon pump
* Carcinoma/major surgery of the pharynx, larynx or esophagus
* Aneurysms of the thoracic aorta
* Tissue necrosis of the esophagus or nasal passage
* Any other medical condition that in the investigator's opinion would render the study procedures dangerous.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 10 individuals aged 18-60 who have sustained an acute traumatic SCI above T2 spinal level less than 72hours prior.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2018-05-16 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
daily resting ejection fraction | up to 3 days
  Index of systolic cardiac function

SECONDARY OUTCOMES:
slope of the Starling curve | up to 3 days
  Slope of the central venous pressure vs. cardiac output curve derived from the fluid challenge

CONTACTS AND LOCATIONS:
Locations (1):
- Vancouver General Hospital, Vancouver, Canada

IPD SHARING:
Plan to Share IPD: No